CLINICAL TRIAL: NCT05533333
Title: Cost-effectiveness of Self-administered Dual-task Training (sDTT) for Reducing Falls Among Older Adults: A Multi-centre-randomized Controlled Trial With Economic Evaluation
Brief Title: Self-administered Dual-task Training for Reducing Falls Among the Older Adults
Acronym: sDTT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other); National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0034640
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-11

CONDITIONS: Older Adults
Keywords: Falls; Older adults; Dual-task; Balance

STUDY DESIGN:
Intervention Model Description: Assessor-blinded, multi-centre parallel-group RCT with economic evaluation
Who Masked: Outcomes Assessor
Masking Description: A person not involved in the study (student helper #1) will randomise the participants using a random number list prepared by Dr Chen Huijun Cynthia (statistician) before the baseline assessment. One HK-registered physiotherapist (RA1) will be recruited to conduct workshops on teaching the exercise interventions to all participants. One research postgraduate (RPg) student will be recruited to conduct all of the other methodological procedures involved in the project. Assessments will be performed by an existing postgraduate student of the PI, who is blind to treatment condition. An economic evaluation with healthcare utility estimation will be performed by Dr Chen Huijun Cynthia. The treatment allocation coding will be unblinded following the completion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self administered dual-task training (Experimental): The exercise intervention will continue for 9 months, beginning with 12 weeks of training accompanied by workshops to teach the exercises.
  Experimental group: sDTT group participants will be instructed to perform 10 minutes of warm-up, 40 minutes of dual-task training and 10 minutes of cool-down exercises. The size of the workshop will be limited to 10 participants. The sDTT programme includes performing a selection of six cognitive tasks during walking, the sit-to-stand movement, heel and toe raising, stepping, tandem standing and walking and multidirectional reaching tasks. The cognitive tasks will include mental tracking, working memory, auditory cues and verbal fluency tasks. Participants will be given the freedom to mix and match the physical and cognitive tasks to make them more challenging.
  Interventions: Behavioral: Falls prevention exercises
- Self-administered singletask training (Active Comparator): Control group: The self-administered single-task training group will receive 10 minutes of warm-up, 20 minutes of physical tasks (as outlined above) and 20 minutes of cognitive tasks (as outlined above) followed by 10 minutes of cool-down exercises. Participants will be instructed to perform the exercises for the same dosage as the experimental group. After a 6-month follow-up period, the control group will receive two complimentary sessions of self-administered dual-task training.
  Interventions: Behavioral: Falls prevention exercises

INTERVENTIONS:
Behavioral: Falls prevention exercises — A dual-task activity involves the simultaneous performance of two activities involving physical and cognitive tasks.
  Other Names: Balance exercises

SUMMARY:
Evidence supports that dual-task training reduces fall risk among older adults. However, the current framework for preventive care for fall prevention in Hong Kong does not include formal cognitive training, while little to no emphasis is placed on combining physical and cognitive training (dual tasking) to prevent falls. Secondly, the healthcare costs for eligible Hong Kong citizens are subsidised by between 81 and 97% of the actual treatment cost. Therefore, there is a demanding need for cost-effective treatment to reduce the country's' economic burden. This project will assist policymakers and clinicians in recommending cost-effective treatments for fall prevention.

DETAILED DESCRIPTION:
Objective: Evaluate the effectiveness and cost-effectiveness of self-administered dual-task training (sDTT) for preventing falls among older adults and promote this technique to the target population and healthcare workers of Hong Kong.

Design: In Phase 1, a multi-centre randomised controlled trial (RCT) with economic evaluation will evaluate the effectiveness and cost-effectiveness. In Phase 2, the technique will be promoted through hands-on workshops for older adults and helpers; and promotional talks with physiotherapists and rehabilitation nurses.

Setting: Community-based elderly care centres. Participants: For the RCT, we will recruit 190 community-dwelling older (≥65 years) adults of both genders having experienced at least one fall in the past 6 months. 500 community-dwelling older adults will be recruited for the workshop and 100 healthcare workers will be engaged for promotion activities.

Intervention: In Phase 1, the experimental group will receive sDTT from a physiotherapist once every 2 weeks for 12 weeks. They will perform home exercises once per week for 12 weeks. Unsupervised exercises will then continue over the next 6 months. Control group will receive the same amount of self-administered single-task training as the experimental group.

Primary outcome measure: Number of falls will be assessed at baseline (T1), post-intervention after 12 weeks (T2) and 6 months (T3). Health promotion will be assessed using a knowledge and attitude questionnaire.

Analysis: General linear mixed model with maximum likelihood estimation will compare primary and secondary outcome measures. Cost-effectiveness will be assessed from the Hong Kong healthcare perspective. Wilcoxon Signed-Rank test will assess the benefits of health promotion.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling
* Ambulant with or without the use of a walking assistive device
* Have experienced at least one fall over the past 6 months and
* Obtained a mini-mental state examination score of ≥ 24 (indicating the absence of cognitive impairment).

Exclusion Criteria:

* Have been diagnosed with dementia or Alzheimer's disease,
* Have a previous history of psychiatric illness
* Are only able to walk with hand-held support
* Have a severe visual impairment that prevents exercise participation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of falls | Change score at week 12 and week 36
  The number of falls will be recorded from the baseline using each participant's digital diary interface. Participants will be instructed to record the number of falls on a weekly basis. The baseline assessment of falls will be calculated as the number of falls over the past 3 months from the day of study enrolment

SECONDARY OUTCOMES:
Dual-task cost of balance performance will be assessed for the TUG | Change score at week 12 and week 36
  Based on the scores of the standard TUG (single task), d-TUG (dual-task TUG) test and standard counting backwards, the dual-task cost of balance performance will be estimated using the formula: (d-TUG - Standard TUG)/ Standard-TUG) × 100.
Dual-task cost of cognitive performance will be assessed for the TUG | Change score at week 12 and week 36
  Based on the scores of the standard TUG (single task), d-TUG (dual-task TUG) test and standard counting backwards, the dual-task cost of balance performance will be estimated using the formula: (d-TUG - Standard counting backwards)/ Standard counting backwards) × 100.
Berg Balance Scale (BBS) | Change score at week 12 and week 36
  The functional balance will be assessed using the 14 item Berg Balance Scale. The Berg Balance Scale has a minimum score of 0 and a maximum of 56 with higher the score better the balance.
Falls Efficacy Scale- International (FES-I) | Change score at week 12 and week 36
  The fear of falls will be assessed using the Falls Efficacy Scale- International (FES-I). This self-reported scale requires the user to rate 16 items between 1 and 4 where 1 implies no difficulty and 4 indicates maximum difficulty. The scale is scored from 16 to 64 with higher the scores indicating higher concerns of falling
12-item Short Form Health Survey (SF-12) | Change score at week 12 and week 36
  The quality of life will be assessed using the 12-item Short Form Health Survey (SF-12) questionnaire. This self-reported questionnaire requires users to complete 12 questions that covers eight domains relevant to general measure of health. An online calculator will be used to derive the final score
Montreal Cognitive Assessment (MoCA) | Change score at week 12 and week 36
  Montreal Cognitive Assessment (MoCA) estimates memory, executive function, attention, language, abstraction, naming, delayed recall and orientation. This brief tool scores cognitive function out of 30, with a higher score equating to better function.
EuroQol 5 dimension 5 level EQ5D5L | Change score at week 12 and week 36
  Health status will be assessed using the EuroQol-5-dimension-5-level (EQ-5D-5L). It is a standardised measure of health status used for economic appraisal. The Chinese translated version of the EQ 5D 5L will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong

REFERENCES:
- [Derived] Khan MJ, Fong KNK, Wong TW, Tsang WW, Chen CH, Chan WC, Winser S. Self-administered dual-task training reduces balance deficits and falls among community-dwelling older adults: a multicentre parallel-group randomised controlled trial with economic evaluation protocol. BMJ Open. 2025 Jun 24;15(6):e089915. doi: 10.1136/bmjopen-2024-089915. PMID 40555445